CLINICAL TRIAL: NCT04557280
Title: A Randomized, Open-label, 3-period Cross-over Study to Assess the Pharmacokinetics of Selatogrel (ACT-246475) in Healthy Subjects After Subcutaneous Administration by Syringe and Auto-injector
Brief Title: A Comparative Study of Selatogrel (ACT-246475) Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ID-076-105
Record Dates: First submitted 2020-09-07; First posted 2020-09-21 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, 3-period crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Treatment A: liquid formulation via auto-injector (Experimental): Selatogrel will be administered as a liquid formulation in a sealed prefilled syringe in an auto-injector forming an integral ready-to-use single-dose drug delivery system.
  Interventions: Combination Product: Selatogrel
- Treatment B: liquid formulation via syringe (Experimental): Selatogrel will be administered as a liquid formulation in a sealed prefilled syringe.
  Interventions: Combination Product: Selatogrel
- Treatment C: lyophilizate-based formulation via syringe (Experimental): Selatogrel will be administered as a reconstituted lyophilizate-based formulation for injection.
  Interventions: Drug: Selatogrel

INTERVENTIONS:
Combination Product: Selatogrel — A single subcutaneous injection of 16 mg.
  Other Names: ACT-246475
  Arms: Treatment A: liquid formulation via auto-injector; Treatment B: liquid formulation via syringe
Drug: Selatogrel — A single subcutaneous injection of 16 mg.
  Other Names: ACT-246475
  Arms: Treatment C: lyophilizate-based formulation via syringe

SUMMARY:
The main purpose is to study the pharmacokinetics of selatogrel (ACT-246475) using different administration modes and formulations. The clinical pharmacology data will be used to support demonstration of bioequivalence and interchangeability of the different formulations.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Healthy male or female participant aged between 18 and 59 years (inclusive) at screening.
* Body mass index of 18.0 to 31.9 kg/m2 (inclusive) at screening and a minimum weight of 50.0 kg at screening and on Day -1.
* Systolic blood pressure 100 to 140 mmHg, diastolic blood pressure 50 to 90 mmHg, and pulse rate 45 to 100 bpm (inclusive), measured on the left arm, after 5 minutes in the supine position at screening and Day-1.
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, measured after 5 min in the supine position at screening and on Day-1.
* Clinical laboratory values are within the standard normal ranges or determined to be clinically insignificant in the opinion of the investigator at screening and on Day -1.
* Women must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline (i.e., Day -1 of the first period). Women of childbearing potential must consistently and correctly use (from screening, during the entire study, and for at least 30 days after last study treatment injection) an acceptable effective method of contraception, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must be initiated at least 1 month before first treatment administration.
* Women of non-childbearing potential.

Exclusion Criteria:

* Pregnant or lactating woman.
* Previous exposure to selatogrel (ACT-246475).
* Previous treatment with acetylsalicylate, non-steroidal anti-inflammatory drugs, P2Y12 receptor antagonists, or any medication with blood-thinning activity (i.e., injectable or oral anticoagulants) within 3 weeks prior to study treatment administration.
* Treatment with another investigational small molecule drug within 30 days or 5 x terminal half-lives ([t½], whichever is longer) or with an investigational biologic drug within 90 days prior to screening.
* Known hypersensitivity to P2Y12 receptor antagonists or to excipients used in any of the formulations.
* History or clinical evidence of alcoholism or drug abuse within 3 years prior to screening.
* History of major medical or surgical disorders, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Family or personal history of prolonged bleeding (e.g., after surgical intervention) or bleeding disorders (e.g., thrombocytopenia, clotting disturbances), intracranial vascular diseases, stroke, transient ischemic attack, reasonable suspicion of vascular malformations, peptic ulcers.
* Platelet count less than 120 x10^9 per litre at screening and on Day-1.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC0-t) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
The area under the plasma concentration-time curve from zero to infinity (AUC0-inf) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
The maximum plasma concentration (Cmax) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Time to reach Cmax (tmax) | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Terminal half-life (t½) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic supine blood pressure | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in pulse rate | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in body weight | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in the electric activity of the heart (12-lead electrocardiogram) | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
  Changes in the PQ-, PR-, RR-, and QRS-interval will be measured. In addition, the QTc-interval corrected for heart rate using Bazett's (QTcB) and Fridericia's formula (QTcF) will be assessed.
Change from baseline in coagulation laboratory tests | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
  Blood samples will be taken under fasted conditions and the following tested: prothrombin time and international normalized ratio, as well as activated partial thromboplastin time.
Change from baseline in clinical chemistry tests | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
  Blood samples will be taken under fasted conditions and the following tested: aspartate aminotransferase / alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, total and direct bilirubin, lactate dehydrogenase; creatinine, urea; urate; glucose; cholesterol, triglycerides; sodium, potassium, chloride, calcium; protein, albumin.
Change from baseline in clinical hematology tests | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
  Blood samples will be taken under fasted conditions and the following tested: hemoglobin, hematocrit, erythrocytes, leukocytes; as well as a differential blood count (including basophils, eosinophils, neutrophils, lymphocytes and monocytes); and platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Altasciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zenklusen I, Hsin CH, Schilling U, Kankam M, Krause A, Ufer M, Dingemanse J. Transition from Syringe to Autoinjector Based on Bridging Pharmacokinetics and Pharmacodynamics of the P2Y12 Receptor Antagonist Selatogrel in Healthy Subjects. Clin Pharmacokinet. 2022 May;61(5):687-695. doi: 10.1007/s40262-021-01097-9. Epub 2021 Dec 28. PMID 34961905